CLINICAL TRIAL: NCT02587325
Title: A Phase 1/1b Clinical Trial of ABI-009, an mTOR Inhibitor, for Patients With Severe Pulmonary Arterial Hypertension (PAH)
Brief Title: Phase 1/1b Study With Nab-sirolimus for Patients With Severe Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aadi Bioscience, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAH-001
Record Dates: First submitted 2015-10-23; First posted 2015-10-27 (Estimated); Results first posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-10

CONDITIONS: Pulmonary Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Nab-Sirolimus Dose Cohort 1 (Experimental): nab-Sirolimus Dose Cohort 1 at 10 mg/m2, given once weekly intravenously for 16 weeks. The initial 16-Week treatment was followed optionally by up to 32 weeks of therapy (Extension Part)
  Interventions: Drug: nab-sirolimus
- Nab-Sirolimus Dose Cohort 2 (Experimental): nab-Sirolimus Dose Cohort 2 at 1.0 mg/m2, given once weekly intravenously for 16 weeks. The initial 16-Week treatment was followed optionally by up to 32 weeks of therapy (Extension Part)
  Interventions: Drug: nab-sirolimus
- Nab-Sirolimus Dose Cohort 3 (Experimental): nab-Sirolimus Dose Cohort 3 at 2.5 mg/m2, given once weekly intravenously for 16 weeks. The initial 16-Week treatment was followed optionally by up to 32 weeks of therapy (Extension Part)
  Interventions: Drug: nab-sirolimus
- Nab-Sirolimus Dose Cohort 4 (Experimental): nab-Sirolimus Dose Cohort 4 at 5.0 mg/m2, given once weekly intravenously for 16 weeks. The initial 16-Week treatment was followed optionally by up to 32 weeks of therapy (Extension Part)
  Interventions: Drug: nab-sirolimus
- Nab-Sirolimus Dose Cohort 5 (Experimental): nab-Sirolimus Dose Cohort 5 at 7.5 mg/m2, given once weekly intravenously for 16 weeks. The initial 16-Week treatment was followed optionally by up to 32 weeks of therapy (Extension Part)
  Interventions: Drug: nab-sirolimus

INTERVENTIONS:
Drug: nab-sirolimus — nab-sirolimus is an mTOR inhibitor
  Other Names: ABI-009, nab-rapamycin

SUMMARY:
mTOR activation has been shown to be relevant in the development and progression of pulmonary hypertension. Inhibition of mTOR has been shown to reverse or regress pulmonary hypertension in animal models. nab-Sirolimus (also known as ABI-009, nab-rapamycin) is an albumin-bound mTOR inhibitor with improved penetration in lung tissue.

DETAILED DESCRIPTION:
nab-Sirolimus, an mTOR inhibitor, is a novel formulation of albumin-bound sirolimus nanoparticles and has produced encouraging results in oncology at doses up to 100 mg/m2 given once weekly IV. This study is aimed to determine the optimal clinial dose of once weekly IV nab-sirolimus in patients with PAH and safety of 16 weeks of therapy (Phase 1, Dose finding Safety Part) followed optionally by up to 32 weeks of therapy (Extension Part).

ELIGIBILITY:
Inclusion Criteria:

* Male or female age >18 years old with a current diagnosis of WHO Group 1 PAH including idiopathic pulmonary arterial hypertension (IPAH), heritable pulmonary arterial hypertension (HPAH), drug and toxin induced PAH, or PAH associated with connective tissue disease, or congenital heart defects (repaired greater than 1 year prior to Screening)
* Must meet following hemodynamic definition prior to initiation of study drug

  * Mean PAP of ≥ 25 mm Hg
  * PCWP or left ventricular end diastolic pressure (LVEDP) of ≤ 15 mm
  * PVR > 5 mmHg/L/min (Woods unit)
* Functional class II or III according to the WHO set forth at the Dana Point Classification 2008 Meeting
* On 2 or more specific standard PAH therapies (for ≥ 8 consecutive weeks and at stable dose for ≥ 4 consecutive weeks) unless documented inability to tolerate 2 standard therapies
* Meet the following criteria determined by pulmonary function tests completed no more than 24 weeks prior to screening, performed with or without bronchodilation:

  * Forced expiratory volume in one second (FEV1) ≥ 55% of predicted normal
  * FEV1:forced vital capacity (FVC) ratio ≥ 0.60
* 6MWD ≥150 meters and ≤450 meters
* Negative serum pregnancy test
* Female of childbearing age either surgically sterilized or using acceptable method of contraception
* Ability to provide written informed consent by the patient or legal guardian

Exclusion criteria:

* History of heart disease including left ventricular ejection fraction (LVEF) ≤ 40% or clinically significant valvular constrictive or atherosclerotic heart disease (myocardial infarction, angina, cerebrovascular accident)
* History of malignancy in 2 years prior to enrollment
* Pulmonary hypertension (PH) belonging to groups 2 to 5 of the 2013 Nice classification
* Current or recent (< 3 months) use of inotropic or vasopressor agents for the treatment of PAH
* Recent (< 2 months) PAH related hospital admission
* History of allergic reactions attributed to compounds of similar chemical or biologic composition including macrolide (eg, azithromycin, clarithromycin, dirithromycin, and erythromycin) and ketolide antibiotics
* Uncontrolled diabetes mellitus as defined by HbA1c >8% despite adequate therapy
* Uncontrolled hyperlipidemia (serum triglyceride ≥300 mg/dL)
* Serum cholesterol ≥350 mg/dL
* Surgery within 3 months of start date of study drug
* Baseline cytopenias:

  * Absolute Neutrophil Count ≤ 1.5 x 109/L
  * Hemoglobin ≤ 9 g/dL
  * Platelet count < 100,000/mm3
* Baseline liver disease: ALT/AST, total bilirubin, alkaline phosphatase >1.5 x ULN
* Baseline renal disease: creatinine >1.5 ULN and/or creatinine clearance (Cockcroft formula) ≤ 30 mL/min
* Inability to attend scheduled clinic visits
* Prior use of study drug within previous 6 months from enrollment
* Previous lung transplant
* Naïve to available standard PAH therapy
* Concomitant genetic or acquired immunosuppressive diseases (such as HIV, AIDS)
* Uncontrolled intercurrent illness that in the opinion of the investigator would limit compliance and tolerance to study requirements (eg, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, diabetes, uncontrolled hypertension, coronary artery disease, or psychiatric illness/social situations)
* Concomitant enrollment in another investigational treatment protocol for PAH
* Use of strong inhibitors and inducers of CYP3A4 within the 14 days prior to receiving the first dose of ABI-009. Additionally, use of any known CYP3A4 substrates with narrow therapeutic window (such as fentanyl, alfentanil, astemizole, cisapride, dihydroergotamine, pimozide, quinidine, terfanide) within the 14 days prior to receiving the first dose of ABI-009

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2022-08-16 (Actual); Study Completion 2022-09-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc Simon, MD, Principal Investigator — University of California, San Francisco
Locations (6):
- United States (6):
  - University of Arizona, Tucson, Arizona
  - Harbor-UCLA Medical Center, Torrance, California
  - Indiana University, Indianapolis, Indiana
  - National Institutes of Health, Bethesda, Maryland
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Inova Fairfax Hospital, Falls Church, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Nab-Sirolimus Dose Cohort 1: nab-Sirolimus Dose Cohort 1 at 10 mg/m^2, given once weekly intravenously for 16 weeks. The initial 16-Week treatment was followed optionally by up to 32 weeks of therapy (Extension Part)
- Nab-Sirolimus Dose Cohort 2: nab-Sirolimus Dose Cohort 2 at 1.0 mg/m^2, given once weekly intravenously for 16 weeks. The initial 16-Week treatment was followed optionally by up to 32 weeks of therapy (Extension Part)
- Nab-Sirolimus Dose Cohort 3: nab-Sirolimus Dose Cohort 3 at 2.5 mg/m^2, given once weekly intravenously for 16 weeks. The initial 16-Week treatment was followed optionally by up to 32 weeks of therapy (Extension Part)
- Nab-Sirolimus Dose Cohort 4: nab-Sirolimus Dose Cohort 4 at 5.0 mg/m^2, given once weekly intravenously for 16 weeks. The initial 16-Week treatment was followed optionally by up to 32 weeks of therapy (Extension Part)
- Nab-Sirolimus Dose Cohort 5: nab-Sirolimus Dose Cohort 5 at 7.5 mg/m^2, given once weekly intravenously for 16 weeks. The initial 16-Week treatment was followed optionally by up to 32 weeks of therapy (Extension Part)
Period: 16-Week Dose-finding Safety Part
Arm/Group | Nab-Sirolimus Dose Cohort 1 | Nab-Sirolimus Dose Cohort 2 | Nab-Sirolimus Dose Cohort 3 | Nab-Sirolimus Dose Cohort 4 | Nab-Sirolimus Dose Cohort 5
Started | 4 | 3 | 4 | 3 | 1
Completed | 3 | 3 | 4 | 2 | 1
Not Completed | 1 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0
Not completed — COVID-19 risk | 0 | 0 | 0 | 1 | 0
Period: 32-Week Optional Extension Part
Arm/Group | Nab-Sirolimus Dose Cohort 1 | Nab-Sirolimus Dose Cohort 2 | Nab-Sirolimus Dose Cohort 3 | Nab-Sirolimus Dose Cohort 4 | Nab-Sirolimus Dose Cohort 5
Started (Optional up to 32-Week Therapy (Extension Part): After the Dose Cohort 1 completed the first 16-Week therapy, the protocol was amended to include an optional up to 32 additional weeks of therapy for patients with clinical evidence of benefit as determined by the site investigator, considering available safety and efficacy outcomes at the Week 17 assessment.) | 0 (Optional up to 32-Week therapy (Extension Part) for patients with clinical evidence of benefit as determined by the site investigator, considering available safety and efficacy outcomes at the Week 17 assessment.) | 1 (Optional up to 32-Week therapy (Extension Part) for patients with clinical evidence of benefit as determined by the site investigator, considering available safety and efficacy outcomes at the Week 17 assessment.) | 4 | 1 (Optional up to 32-Week therapy (Extension Part) for patients with clinical evidence of benefit as determined by the site investigator, considering available safety and efficacy outcomes at the Week 17 assessment.) | 1
Completed (The "Optional up to 32-Week therapy (Extension Part)" was a therapy maintenance opportunity as long as clinically/medically indicated per the treating physician.) | 0 | 1 | 2 | 1 | 0
Not Completed | 0 | 0 | 2 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety analysis set includes all treated patients
Groups:
- Nab-Sirolimus Dose Cohort 1: nab-Sirolimus Dose Cohort 1 at 10 mg/m^2, given once weekly intravenously for 16 weeks.
- Nab-Sirolimus Dose Cohort 2: nab-Sirolimus Dose Cohort 2 at 1.0 mg/m^2, given once weekly intravenously for 16 weeks.
- Nab-Sirolimus Dose Cohort 3: nab-Sirolimus Dose Cohort 3 at 2.5 mg/m^2, given once weekly intravenously for 16 weeks.
- Nab-Sirolimus Dose Cohort 4: nab-Sirolimus Dose Cohort 4 at 5.0 mg/m^2, given once weekly intravenously for 16 weeks.
- Nab-Sirolimus Dose Cohort 5: nab-Sirolimus Dose Cohort 5 at 7.5 mg/m^2, given once weekly intravenously for 16 weeks.
- Total: Total of all reporting groups
Arm/Group | Nab-Sirolimus Dose Cohort 1 | Nab-Sirolimus Dose Cohort 2 | Nab-Sirolimus Dose Cohort 3 | Nab-Sirolimus Dose Cohort 4 | Nab-Sirolimus Dose Cohort 5 | Total
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 1 | 15
Age, Continuous [Median (Full Range); unit: years] | 56.5 [52 to 69] | 45 [44 to 63] | 38.5 [20 to 67] | 45 [44 to 67] | 28 [28 to 28] | 45 [20 to 69]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 15 Patients in the 16-week Dose-Finding Safety Part and 7 continued into the 32-Week Optional Extension Part
  Participants
    16-Week Dose-finding Safety Part: Female | 3 | 3 | 4 | 3 | 1 | 14
    16-Week Dose-finding Safety Part: Male | 1 | 0 | 0 | 0 | 0 | 1
    32-Week Optional Extension Part: number analyzed (Participants) | 0 | 1 | 4 | 1 | 1 | 7
    32-Week Optional Extension Part: Female | 0 | 1 | 4 | 1 | 1 | 7
    32-Week Optional Extension Part: Male | 0 | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: 15 patients in the 16-week dose finding part and 7 patients continued to the 32-week optional extension part.
  Participants
    16-Week Dose-finding Safety Part: Hispanic or Latino | 0 | 1 | 1 | 1 | 0 | 3
    16-Week Dose-finding Safety Part: Not Hispanic or Latino | 4 | 2 | 3 | 2 | 1 | 12
    16-Week Dose-finding Safety Part: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
    32-Week Optional Extension Part: number analyzed (Participants) | 0 | 1 | 4 | 1 | 1 | 7
    32-Week Optional Extension Part: Hispanic or Latino | 0 | 1 | 2 | 0 | 0 | 3
    32-Week Optional Extension Part: Not Hispanic or Latino | 0 | 0 | 2 | 1 | 1 | 4
    32-Week Optional Extension Part: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 15 Patients in the 16-week Dose-Finding Safety Part and 7 continued into the 32-Week Optional Extension Part
  Participants
    16-Week Dose-finding Part: American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 1
    16-Week Dose-finding Part: Asian | 0 | 0 | 0 | 0 | 0 | 0
    16-Week Dose-finding Part: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    16-Week Dose-finding Part: Black or African American | 0 | 0 | 0 | 0 | 0 | 0
    16-Week Dose-finding Part: White | 4 | 3 | 3 | 3 | 1 | 14
    16-Week Dose-finding Part: More than one race | 0 | 0 | 0 | 0 | 0 | 0
    16-Week Dose-finding Part: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
    32-Week Optional Extension Part: number analyzed (Participants) | 0 | 1 | 4 | 1 | 1 | 7
    32-Week Optional Extension Part: American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 1
    32-Week Optional Extension Part: Asian | 0 | 0 | 0 | 0 | 0 | 0
    32-Week Optional Extension Part: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    32-Week Optional Extension Part: Black or African American | 0 | 0 | 0 | 0 | 0 | 0
    32-Week Optional Extension Part: White | 0 | 1 | 3 | 1 | 1 | 6
    32-Week Optional Extension Part: More than one race | 0 | 0 | 0 | 0 | 0 | 0
    32-Week Optional Extension Part: Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 4 | 3 | 1 | 15
Body Surface Area [Median (Full Range); unit: m^2] — Population: 15 Patients in the 16-week Dose-Finding Safety Part and 7 continued into the 32-Week Optional Extension Part
  m^2
    16-Week Dose-finding Safety Part | 2.1 [1.5 to 2.5] | 1.6 [1.5 to 1.7] | 1.6 [1.5 to 1.9] | 1.8 [1.5 to 1.9] | 1.8 [1.8 to 1.8] | 1.7 [1.5 to 2.5]
    32-Week Optional Extension Part: number analyzed (Participants) | 0 | 1 | 4 | 1 | 1 | 7
    32-Week Optional Extension Part |  | 1.5 [1.5 to 1.5] | 1.7 [1.5 to 1.9] | 1.9 [1.9 to 1.9] | 1.8 [1.8 to 1.8] | 1.8 [1.5 to 1.9]

OUTCOME MEASURES:

1. Primary Outcome: Dose-limiting Toxicities
Description: A dose-limiting toxicity (DLT) was defined as a study drug-related Grade ≥3 hematologic AE or persistent intolerable nonhematologic AE of any grade that occurred during the first 4 weeks of treatment, requiring dose reduction or permanent discontinuation of the study drug, in the opinion of the Investigator. The number and percent of patients with a DLT were to be reported by dose cohorts in the Phase 1 dose finding part of the study if any were observed in the study.
Time Frame: 16 weeks
Population: The Treated Population included all patients who received at least 1 dose of nab sirolimus. This population was used for analyses of safety.
Measure: Count of Participants; unit: Participants
Arm/Group | Nab-Sirolimus Dose Cohort 1 | Nab-Sirolimus Dose Cohort 2 | Nab-Sirolimus Dose Cohort 3 | Nab-Sirolimus Dose Cohort 4 | Nab-Sirolimus Dose Cohort 5
Number analyzed (Participants) | 4 | 3 | 4 | 3 | 1
Participants | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Right Heart Catheterization Based on Central Lab Analysis (Pulmonary Vascular Resistance, Cardiac Output, Cardiac Index, Stroke Volume)
Description: Median Percent Change from Baseline to Week 17 (after 16 weeks of treatment) in RHC based on Central Lab Analysis (Pulmonary vascular resistance, Cardiac Output, Cardiac Index, Stroke Volume)
Time Frame: 17 Weeks
Population: The Efficacy Evaluable Population included all patients who received at least 1 dose of nab-sirolimus and had at least one post-baseline efficacy assessment. This population was used for analyses of efficacy (N=13).
Measure: Median (Full Range); unit: percentage of change
Groups:
- Overall: nab-Sirolimus Dose Cohort 1-5 at 1-10 mg/m2, given once weekly intravenously for 16 weeks. The initial 16-Week treatment was followed optionally by up to 32 weeks of therapy (Extension Part).
Arm/Group | Nab-Sirolimus Dose Cohort 1 | Nab-Sirolimus Dose Cohort 2 | Nab-Sirolimus Dose Cohort 3 | Nab-Sirolimus Dose Cohort 4 | Nab-Sirolimus Dose Cohort 5 | Overall
Number analyzed (Participants) | 3 | 3 | 4 | 2 | 1 | 13
percentage of change
  Pulmonary Vascular Resistance (dyn×sec/cm5) | -30.1 [-47.8 to -21.8] | 10.9 [-20.5 to 18.0] | -3.5 [-40.2 to 14.5] | -15.7 [-33.3 to 1.9] | -30.8 [-30.8 to -30.8] | -20.5 [-47.8 to 18.0]
  Thermodilution Cardiac Output Mean (L/minute) | 40.1 [39.5 to 59.6] | -15.4 [-23.1 to -13.1] | 10.8 [-15.6 to 40.1] | 9.6 [-9.4 to 28.5] | 27.4 [27.4 to 27.4] | 16.9 [-23.1 to 59.6]
  Cardiac Index (L/minute/m2) | 40.1 [39.5 to 66.4] | -16.5 [-17.4 to -12.8] | 13.5 [-17.2 to 43.9] | 9.4 [-5.7 to 24.5] | 31.2 [31.2 to 31.2] | 21.4 [-17.4 to 66.4]
  Stroke Volume (mL) | 11.6 [11.1 to 81.1] | -14.4 [-19.4 to 10.3] | 11.0 [-24.6 to 42.3] | 6.3 [-14.6 to 27.1] | 10.5 [10.5 to 10.5] | 10.5 [-24.6 to 81.1]

3. Secondary Outcome: 6-minute Walk Distance (6MWD)
Description: Median Percent Change from Baseline to Week 17 (after 16 weeks of treatment) in 6MWD
Time Frame: 17 Weeks
Population: as for outcome 2
Measure: Median (Full Range); unit: percentage of change
Arm/Group | Nab-Sirolimus Dose Cohort 1 | Nab-Sirolimus Dose Cohort 2 | Nab-Sirolimus Dose Cohort 3 | Nab-Sirolimus Dose Cohort 4 | Nab-Sirolimus Dose Cohort 5 | Overall
Number analyzed (Participants) | 3 | 3 | 4 | 2 | 1 | 13
percentage of change | -2.0 [-21.0 to 46.6] | 16.0 [3.1 to 37.8] | 13.3 [-14.0 to 22.5] | 16.6 [12.3 to 21.0] | 21.0 [21.0 to 21.0] | 15.0 [-21.0 to 46.6]

4. Secondary Outcome: N-terminal Pro-brain Natriuretic Peptide (NT Pro-BNP)
Description: Median Percent Change from Baseline to Week 17 (after 16 weeks of treatment) in NT Pro-BNP
Time Frame: 17 Weeks
Population: The Efficacy Evaluable Population included all patients who received at least 1 dose of nab-sirolimus and had at least one post-baseline efficacy assessment. This population was used for analyses of efficacy (N=12).
Measure: Median (Full Range); unit: percentage of change
Arm/Group | Nab-Sirolimus Dose Cohort 1 | Nab-Sirolimus Dose Cohort 2 | Nab-Sirolimus Dose Cohort 3 | Nab-Sirolimus Dose Cohort 4 | Nab-Sirolimus Dose Cohort 5 | Overall
Number analyzed (Participants) | 3 | 3 | 3 | 2 | 1 | 12
percentage of change | -49.0 [-65.5 to 79.7] | -34.6 [-73.8 to -4.5] | -7.1 [-62.2 to 18.8] | -10.8 [-21.6 to 0.0] | -17.0 [-17.0 to -17.0] | -19.3 [-73.8 to 79.7]

ADVERSE EVENTS:
Time Frame: Adverse Events reported in the initial 16-Week Treatment for all Cohorts 1,2,3,4 & 5 (ie, from baseline through Week 16). Adverse Events reported in the Optional Extension Phase for up to additional 32 weeks of treatment for Cohorts 2, 3, 4, and 5 (ie, Week 17 through 48).
Groups:
- Nab-Sirolimus Dose Cohort 1: nab-Sirolimus Dose Cohort 1 at 10 mg/m2, given once weekly intravenously for 16 weeks.
- Nab-Sirolimus Dose Cohort 2: nab-Sirolimus Dose Cohort 2 at 1.0 mg/m2, given once weekly intravenously for 16 weeks.
- Nab-Sirolimus Dose Cohort 3: nab-Sirolimus Dose Cohort 3 at 2.5 mg/m2, given once weekly intravenously for 16 weeks.
- Nab-Sirolimus Dose Cohort 4: nab-Sirolimus Dose Cohort 4 at 5.0 mg/m2, given once weekly intravenously for 16 weeks.
- Nab-Sirolimus Dose Cohort 5: nab-Sirolimus Dose Cohort 5 at 7.5 mg/m2, given once weekly intravenously for 16 weeks.
- Overall Nab-Sirolimus Dose Cohort 1-5: nab-Sirolimus Dose Cohort 1-5 at 1-10 mg/m2, given once weekly intravenously for 16 weeks.
- Nab-Sirolimus Dose Cohort 2; 32 Weeks Optional Extension: The initial 16-Week treatment at 1.0 mg/m2 was followed optionally by up to 32 weeks of therapy (Extension Part)
- Nab-Sirolimus Dose Cohort 3; 32 Weeks Optional Extension: The initial 16-Week treatment at 2.5 mg/m2 was followed optionally by up to 32 weeks of therapy (Extension Part)
- Nab-Sirolimus Dose Cohort 4; 32 Weeks Optional Extension; Nab-Sirolimus Dose Cohort 5; 32 Weeks Optional Extension: The initial 16-Week treatment at 5.0 mg/m2 was followed optionally by up to 32 weeks of therapy (Extension Part)
Arm/Group | Nab-Sirolimus Dose Cohort 1 | Nab-Sirolimus Dose Cohort 2 | Nab-Sirolimus Dose Cohort 3 | Nab-Sirolimus Dose Cohort 4 | Nab-Sirolimus Dose Cohort 5 | Overall Nab-Sirolimus Dose Cohort 1-5 | Nab-Sirolimus Dose Cohort 2; 32 Weeks Optional Extension | Nab-Sirolimus Dose Cohort 3; 32 Weeks Optional Extension | Nab-Sirolimus Dose Cohort 4; 32 Weeks Optional Extension | Nab-Sirolimus Dose Cohort 5; 32 Weeks Optional Extension
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 0/4 | 0/3 | 0/1 | 0/15 | 0/1 | 0/4 | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 1/4 | 0/3 | 0/4 | 1/3 | 0/1 | 2/15 | 0/1 | 1/4 | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 4/4 | 3/3 | 1/1 | 15/15 | 0/1 | 4/4 | 1/1 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nab-Sirolimus Dose Cohort 1 (N=4) | Nab-Sirolimus Dose Cohort 2 (N=3) | Nab-Sirolimus Dose Cohort 3 (N=4) | Nab-Sirolimus Dose Cohort 4 (N=3) | Nab-Sirolimus Dose Cohort 5 (N=1) | Overall Nab-Sirolimus Dose Cohort 1-5 (N=15) | Nab-Sirolimus Dose Cohort 2; 32 Weeks Optional Extension (N=1) | Nab-Sirolimus Dose Cohort 3; 32 Weeks Optional Extension (N=4) | Nab-Sirolimus Dose Cohort 4; 32 Weeks Optional Extension (N=1) | Nab-Sirolimus Dose Cohort 5; 32 Weeks Optional Extension (N=1)
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Device Related Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nab-Sirolimus Dose Cohort 1 (N=4) | Nab-Sirolimus Dose Cohort 2 (N=3) | Nab-Sirolimus Dose Cohort 3 (N=4) | Nab-Sirolimus Dose Cohort 4 (N=3) | Nab-Sirolimus Dose Cohort 5 (N=1) | Overall Nab-Sirolimus Dose Cohort 1-5 (N=15) | Nab-Sirolimus Dose Cohort 2; 32 Weeks Optional Extension (N=1) | Nab-Sirolimus Dose Cohort 3; 32 Weeks Optional Extension (N=4) | Nab-Sirolimus Dose Cohort 4; 32 Weeks Optional Extension (N=1) | Nab-Sirolimus Dose Cohort 5; 32 Weeks Optional Extension (N=1)
Diarrhea (Gastrointestinal disorders) | 3 | 1 | 1 | 2 | 0 | 7 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 1 | 0 | 3 | 1 | 7 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 3 | 1 | 2 | 1 | 9 | 0 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 2 | 1 | 7 | 0 | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 1 | 3 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 1 | 2 | 0 | 5 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 3 | 0 | 3 | 0 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 0 | 1 | 4 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0 | 3 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 0 | 3 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 1 | 0 | 5 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 0 | 3 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Myelosuppression (Thrombocytopenia) (Blood and lymphatic system disorders) | 2 | 1 | 1 | 0 | 0 | 4 | 0 | 0 | 0 | 0
Mucositis (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Dry Mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Lip Blister (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The originally planned dose levels started at 10 mg/m2 weekly nab-sirolimus. While there were no DLTs at the initial dose level (n = 4), based on the totality of AEs and dose reductions, dose levels were modified and patients sequentially enrolled at 1.0, 2.5, 5.0, and 7.5 mg/m2. Given the difficulties with enrollment during the COVID-19 pandemic, the study closed prior to fully enrolling at the last dose level of 7.5 mg/m2 and thus, no Phase 1b cohort expansion occurred at this dose.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-24): https://cdn.clinicaltrials.gov/large-docs/25/NCT02587325/Prot_SAP_000.pdf